CLINICAL TRIAL: NCT00974610
Title: Collaborative Project on Potential Serum Markers for Malignant Melanoma, Metastatic Breast, Advanced Lung Pancreatic Carcinoma and Colorectal Cancer
Brief Title: Study of Blood Samples From Patients With Malignant Melanoma, Metastatic Breast Cancer, Advanced Lung Cancer, Pancreatic Cancer, or Colorectal Cancer.
Status: Completed | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: CTRIAL-IE (ICORG) 07-12; CTRIAL-IE (ICORG) 07-12; EU-20949
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Melanoma (Skin); Pancreatic Cancer
Keywords: stage IV melanoma; recurrent melanoma; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; stage IV breast cancer; recurrent breast cancer; male breast cancer; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent pancreatic cancer; stage IV colon cancer; recurrent colon cancer; stage IV rectal cancer; recurrent rectal cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Melanoma; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Breast Neoplasms, Male; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (5):
- Breast
- Lung
- Melanoma
- Pancreatic
- Colorectal

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in peptides and proteins and identify biomarkers related to cancer.

PURPOSE: This research study is looking at blood samples from patients with malignant melanoma, metastatic breast cancer, advanced lung cancer, pancreatic cancer, or colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess which potential peptide and protein markers produced by human melanoma, lung, breast, pancreatic, and colorectal cell lines may be detectable in serum of patients from these five disease groups.

Secondary

* To conduct further extensive investigation with respect to identification of the protein/peptide involved, determination of specificity for each cancer, and development of more sensitive assays to look for such markers in a wider population of patients, including those undergoing therapy.

OUTLINE: This is a multicenter study.

Blood samples are collected before surgical intervention or treatment to assess peptide and protein markers.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following advanced metastatic malignancies:

  * Malignant melanoma
  * Lung cancer
  * Breast cancer
  * Pancreatic carcinoma
  * Colorectal cancer
* Advanced and/or metastatic disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 5 different tumour types
Sampling Method: Probability Sample
Enrollment: 803 (Actual)
Dates: Start 2008-08; Primary Completion 2015-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Detection of peptide and protein markers in serum | Ongoing

SECONDARY OUTCOMES:
Identification of the protein/peptide involved | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Martin Clynes, Principal Investigator — National Institute for Cellular Biotechnology at Dublin City University
Locations (13):
- Ireland (13):
  - Cork University Hospital, Cork
  - Mercy University Hospital, Cork
  - Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St Luke's Hospital, Dublin
  - University College Hospital, Galway
  - Letterkenny General Hospital, Letterkenny
  - Mid-Western Cancer Centre at Mid-Western Regional Hospital, Limerick
  - Waterford Regional Hospital, Waterford